CLINICAL TRIAL: NCT07407634
Title: Evaluation of XTYW007 in Healthy Subjects and Healthy Subjects With Elevated LDL-C:A Randomized, Double-Blind, Single-Center Phase I/IIa Study of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect Following Single and Multiple Doses
Brief Title: A Randomized, Double-blind, Single-center Phase I/IIa Study of XTYW007 Tablets in Subjects.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Xi'an Xintong Pharmaceutical Research Co.,Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XTYW007-2025-01
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose group (Experimental): Group 1 (0.2 mg), Group 2 (0.6 mg), Group 3 (1.5 mg), Group 4 (3 mg), Group 5, Group A (6 mg), Group 6 (10 mg), Group 7 (15 mg), optional dose Group 8 (20 mg)
  Interventions: Drug: Test drug XTYW007 capsules and placebo,Single dose group
- Food Impact Group (Experimental): Group 5, Subgroup A（6mg）, Group 5, Subgroup B（ 6 mg）
  Interventions: Drug: Test drug XTYW007 capsules and placebo,Food Impact Group
- Multiple dosing group (Experimental): Group 9 (1.5 mg), Group 10 (6 mg), Group 11 (15 mg)
  Interventions: Drug: Test drug XTYW007 capsules and placebo,Multiple dosing group

INTERVENTIONS:
Drug: Test drug XTYW007 capsules and placebo,Single dose group — Each group consists of 8 people, with 6 receiving the trial drug XTYW007 and 2 receiving a placebo. The sentinel method is used for enrollment, meaning that the first 2 subjects (one male and one female, both receiving the trial drug) are enrolled and observed for 96 hours (after the Day 5 tolerance assessment). If there are no intolerable reactions, the remaining 6 subjects are enrolled and randomly assigned to receive the trial drug or placebo in a 2:1 ratio.
  Arms: Single dose group
Drug: Test drug XTYW007 capsules and placebo,Food Impact Group — A two-period crossover administration was used, with a 14-day washout period. In Group A, 8 subjects received the drug on D1 under fasting conditions in the first period, and on D15 under fed conditions in the second period. In Group B, 6 subjects taking the investigational drug received it on D1 under fed conditions in the first period, and on D15 under fasting conditions in the second period.
  Arms: Food Impact Group
Drug: Test drug XTYW007 capsules and placebo,Multiple dosing group — Each group consists of 8 subjects, with 6 receiving the investigational drug XTYW007 and 2 receiving a placebo. A sentinel dosing approach is used, where 2 subjects (one male and one female) are first enrolled and administered the investigational drug. After 96 hours of observation (tolerance evaluation on Day 5), if no intolerable issues occur, the remaining 6 subjects are enrolled and randomized 2:1 to receive the investigational drug or placebo. In the multiple-dose group, the drug is administered once every morning on an empty stomach (QD) for 14 consecutive days.
  Arms: Multiple dosing group

SUMMARY:
Aimed at evaluating the safety, tolerability, and pharmacokinetic characteristics of single and multiple doses of XTYW007 in healthy subjects and healthy subjects with elevated LDL-C, as well as studying the effects of food on the pharmacokinetics and metabolic transformation of XTYW007, and preliminarily assessing the pharmacodynamics of XTYW007.

DETAILED DESCRIPTION:
This study is a single-center, randomized, double-blind Phase I/IIa clinical trial assessing the safety, tolerability, and pharmacokinetics of single and multiple doses.Aimed at evaluating the safety, tolerability, and pharmacokinetic characteristics of single and multiple doses of XTYW007 in healthy subjects and healthy subjects with elevated LDL-C, as well as studying the effects of food on the pharmacokinetics and metabolic transformation of XTYW007, and preliminarily assessing the pharmacodynamics of XTYW007.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily sign the informed consent before the trial, and fully understand the content, process and possible adverse effects of the trial;
2. They are able to complete the study according to the requirements of the trial protocol;
3. Subjects (including partners) are willing to have no pregnancy plan and voluntarily use effective contraceptive measures within 6 months from screening to the last dose of study drug;
4. Male and female subjects between the ages of 18 and 65 (including borderline values);
5. Male subjects weighing not less than 50 kg and female subjects weighing not less than 45 kg. Body mass index (BMI) = weight (kg)/ height 2 (m2), BMI within the range of 18-28 kg/m2 (including the threshold value);
6. During screening, for single-dose studies, fasting low-density lipoprotein cholesterol (LDL-C): 80 mg/dL < LDL-C < 120 mg/dL (2.06 mmol/L ~ 3.1 mmol/L); for multiple-dose studies, fasting low-density lipoprotein cholesterol (LDL-C) > 110 mg/dL (2.85 mmol/L);
7. Physical examination and vital signs are normal or abnormal without clinical significance.

Exclusion Criteria:

1. Individuals with allergic constitution (allergic to multiple drugs and foods) or intolerance to β-blockers;
2. History of thyroid-related diseases and/or thyroid function abnormalities during the screening phase that are clinically significant;
3. Individuals who smoked more than 5 cigarettes per day in the 3 months prior to the trial;
4. History of drug abuse and/or alcoholism (consuming 14 units of alcohol per week: 1 unit = 285 mL beer, 25 mL spirits, or 100 mL wine);
5. Blood donation or significant blood loss (>450 mL) within 3 months prior to taking the study drug;
6. Use of any prescription drugs, over-the-counter drugs, vitamins, herbal products, or alcohol within 14 days before taking the study drug;
7. Consumption of special foods (such as grapefruit, mango, dragon fruit, grape juice, orange juice, etc., rich in flavonoids or coumarins) within 2 weeks before taking the study drug, or engaging in intense exercise, or other factors affecting drug absorption, distribution, metabolism, or excretion;
8. Significant changes in diet or exercise habits recently;
9. Use of the study drug or participation in a drug clinical trial within 3 months before taking the study drug;
10. Difficulty swallowing or any gastrointestinal diseases affecting drug absorption within 6 months prior to the study;
11. Any disease that increases bleeding risk, such as hemorrhoids, acute gastritis, or gastroduodenal ulcer;
12. Clinically significant ECG abnormalities; QTcF > 470 ms (QTcF = QT/(RR)^0.33);
13. Female subjects who are breastfeeding during the screening or trial phase, planning pregnancy in the near future, or have positive serum pregnancy results;
14. Abnormal clinical laboratory test results with clinical significance, or other clinical findings within 12 months prior to screening that are clinically significant, including but not limited to diseases of the gastrointestinal tract, kidney, liver, nervous system, hematopoietic system, endocrine system, tumors, lungs, immune system, mental health, or cardiovascular and cerebrovascular systems;
15. Any positive result for hepatitis B surface antigen, hepatitis C antibody/core antigen, HIV antigen/antibody, or syphilis treponema antibody during screening;
16. Occurrence of acute illness or concomitant medication use from the screening phase to the start of study medication;
17. Consumption of chocolate, any caffeine-containing or xanthine-containing foods or beverages within 24 hours before taking the study drug;
18. Serum creatinine clearance ≤ 70 mL/min [calculation formula: Ccr: (140 - age) × weight (kg) / (0.818 × Scr) (μmol/L), ×0.85 for females];
19. Subjects with special dietary requirements who cannot consume the complete study meal or who do not agree to adhere to water intake regimen and position restrictions during the trial;
20. Subjects whom the investigator considers to have other factors that make them unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2026-03-25 (Estimated); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events | Days 1-11 of administration
  Number of participants who experienced treatment-related adverse events as assessed by CTCAE v5.0.
Cmax | Days 1-11 of administration
  Cmax
Tmax | Days 1-11 of administration
  Tmax
t1/2 | Days 1-11 of administration
  t1/2
AUC | Days 1-11 of administration
  AUC
CL/F | Days 1-11 of administration
  CL/F
Vz/F | Days 1-11 of administration
  Vz/F
CLr/F | Days 1-11 of administration
  CLr/F

SECONDARY OUTCOMES:
Ae0-72 h | Days 1-4 of administration
  Ae0-72 h
Fe0-72 h | Days 1-4 of administration
  Fe0-72 h
Blood lipids | Days 1-11 of administration
  TC , TG , LDL-C, HDL-C, Apo A1, Apo B, Lp(a)
Thyroid function | Days 1-11 of administration
  TSH, TT4, TT3, FT4, FT3
Sex hormone-binding globulin (SHBG) | Days 1-11 of administration
  SHBG

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China